CLINICAL TRIAL: NCT04438538
Title: Risk Factors for the Development of Bilateral Ménière's Disease and the Establishment of a National Ménière's Disease Registry.
Brief Title: Ménière's Disease Registry
Acronym: MDR
Status: Completed | Type: Observational
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other); Ménière's Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: 275749
Record Dates: First submitted 2020-02-26; First posted 2020-06-19 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-07

CONDITIONS: Ménière's Disease
Keywords: patient reported questionnaires; audiometric; vestibular; radiological tests
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Dizziness: All trial participants are within this group. All trial participants will either have a diagnosis or a suspected diagnosis of Ménière's Disease in order to take part.

SUMMARY:
Recent research has suggested that Ménière's disease may be a consequence of a number of individual conditions rather than developing from a single cause. This means that determining the different conditions that cause Ménière's disease will help the investigators to provide effective treatments. Experience from other similar medical conditions has taught the investigators that the best method to identify different causes of a condition is via a process called 'clinical subtyping'.

The investigators intend to set up a large Ménière's disease database in order to allow then to subtype Ménière's disease. More specifically, the proposed project aspires to achieve two aims. The investigators intend to investigate a sub-type of Ménière's disease, bilateral disease, i.e. both ears affected. The study hopes to identify what features predict an individual developing bilateral Ménière's disease. Secondly, to test the feasibility of expanding the database across the whole of the UK to involve all Ménière's disease patients. This will allow many other features of Ménière's disease to be used to establish sub-types and help predict the best treatment for individual patients.

DETAILED DESCRIPTION:
Ménière's disease is an inner ear disorder characterised by recurrent episodes of spontaneous vertigo, fluctuating hearing loss and tinnitus, often with a feeling of fullness in the ear. The exact aetiology remains unknown. Ménière's disease is estimated to have a prevalence of 0.25% in the UK (around 162,000 individuals) (Tyrrell 2016) and is associated with significant physical, psychological and socioeconomic morbidity (Anderson 2001, Tyrrell 2014).

There is a substantial lack of knowledge regarding many aspects of Ménière's disease, including a fuller understanding of epidemiological aspects of the disease, aetiological factors, pathogenesis, clinical course and treatment outcomes. The James Lind Alliance cites Ménière's disease as the theme for four of their top ten priorities for addressing uncertainties in the field of balance disorders (JLA 2018).

There is mounting unease regarding the definition of Ménière's disease as a single clinical entity. Many consider it to represent the final pathway of a number of individual disease processes. This is reflected by the progressive and varied development of diagnostic criteria over the last few decades (Gurkov 2016). It is in the context of these observations that Ménière's disease is likely to represent a heterogeneous clinical condition defined only by small groups of common, but not always mandatory, symptoms. Understanding how Ménière's disease may exist as a cluster of clinical sub-types is key to allowing further research into its underlying pathophysiological mechanisms, and the targeting of specific treatment strategies; as well as allowing a better understanding of the physiology of the inner ear micro-environment (Phillips 2018).

This project will provide the initial steps necessary to set-up a UK Ménière's disease registry by primarily investigating a single clinical subtype of Ménière's disease: bilateral disease. The development of bilateral Ménière's disease has significant implications for short and long-term opportunities for treatment and rehabilitation; this in turn has significant implications for communication and employment. Previous literature on bilateral disease has offered widely ranging estimates of the likelihood that it will occur in cases where unilateral disease is confirmed, and no clear predictors have been identified (Huppert 2010). However, it is a sub-type which is relatively well-defined with standard internationally agreed criteria for diagnosis.

In areas of research such as this, the implementation of bespoke data collection platforms and national registries have been demonstrated to be both effective and efficient (Mandavia 2017). The use of national registries has many advantages over conventional data collection methods. When implemented correctly, national registries can allow the appraisal of a more representative sample of the target population. Furthermore, a national approach broadens the opportunities both for participation among the patient population to be served by such a venture, and for public engagement and dissemination activities.

A national registry would allow the identification of features at presentation that predict disease course and long-term outcome, improving the understanding of disease progression, treatment response, and underlying aetiology. A UK Ménière's disease registry would also provide a resource for broad and far reaching research into Ménière's disease beyond that of defining clinical sub-types. Registries offer other benefits to patients, carers (including partners and family), researchers, clinicians and other individuals that are involved with the provision of services for those affected by the condition being studied. Individual hospitals and the NHS as a whole can use registry data to improve the services they offer. Individual patients and carers can use registries to learn more about their condition and this can lead to a better understanding of how people's lives are affected. It is anticipated that this work will lead to further registry development and expansion with a broad remit of aims via further awards from major research funders.

To develop the methods and infrastructure for a national registry by recruiting participants from three distinct urban and rural regions within the UK (Norfolk, Leicestershire and London). This will include an appraisal of a number of practical processes of recruitment, such as data acquisition, data processing and data management. This will inform future stages to expand the infrastructure to support a registry for widespread national use.

This project will require the retrospective collection of data from existing Ménière's patients.

Potential participants with a diagnosis of probable or definite unilateral or bilateral Ménière's Disease as defined by the 2015 edition of the American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS) criteria (Goebel 2016) in their hospital records will be identified at ENT secondary care and private clinics. Potential participants must have received a diagnosis of Ménière's Disease within the previous 10 years or have received a new diagnosis during the recruitment window of the study. Unilateral and bilateral Ménière's disease will be defined as follows:

Unilateral Ménière's Disease

At least two episodes of vertigo each lasting at least 20 minutes, where each episode is associated with aural symptoms in a single ear.

Bilateral Ménière's Disease

At least two episodes of vertigo each lasting at least 20 minutes, where each episode is associated with aural symptoms in both ears.

Data will include contemporaneous and historical information regarding medical and relevant social/occupational history, audiometric data, vestibular testing data, radiological data and symptom specific and health related quality of life questionnaires. Clinical data will be requested, collected and extracted locally and entered directly into the Study Dataset managed by Norwich Clinical Trials Unit at the University of East Anglia.

Participants will be offered the option of completing the study questionnaires online or on paper (for entry by a member of the research team). No additional outpatient appointments outside normal care pathways will be required.

The full dataset will be composed of three components:

1. Medical history. This will be completed by the participant onto a predefined data collection form - see additional document: MDR_NVPQ
2. Symptom questionnaires. These will be completed by the participant
3. Audiometric, Vestibular and Radiological test results. This will be completed by the local investigator team.

The investigators anticipate that participants will spend no longer than 60 minutes to complete the necessary forms and questionnaires.

Participants will be asked to complete a non-validated Ménière's disease questionnaire about their Ménière's disease including demographics, history, symptoms including triggers of Ménière's disease related vertigo attacks, comorbidities, current treatment and past treatments tried for Ménière's disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over.
* A probable or definite diagnosis of unilateral or bilateral Meniere's disease as defined by the 2015 edition of the American Academy of Otolaryngology-Head and Neck Surgery (Goebel 2016)
* A willingness to provide consent for data from health records to be used for research purposes.

Exclusion Criteria:

* Unable to provide consent
* Unable/unwilling to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or over with a definite or probable diagnosis of Ménière's disease. These will be collated from NHS hospitals and the corresponding clinician's private clinics.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To acquire data on existing Ménière's disease patients from three UK regions. | 20 minutes
  Participants will be asked to complete a non-validated Ménière's disease questionnaire about their Ménière's disease including demographics, history, symptoms including triggers of Ménière's disease related vertigo attacks, comorbidities, current treatment and past treatments tried for Ménière's disease
An estimation of the prevalence and incidence of bilateral disease: | through study completion, an average of 1 year
  The investigators should identify candidate risk factors that would increase or decrease the chances of developing bilateral disease. These could be further tested in a study of incident (i.e. newly occurring) cases of Ménière's disease followed prospectively in time. However, the initial set of risk factors should allow us to start the process of characterising the bilateral subtype and further understanding it aetiology.
Putative risk factors for the conversion from unilateral to bilateral disease: | through study completion, an average of 1 year
  The proportion of individuals with unilateral Ménière's disease that develop bilateral Ménière's disease after defined periods of time. Ultimately, it would be useful if the investigators could inform patients that, for example, if they haven't developed bilateral disease after a defined number of years from referral to secondary care, their chance of developing bilateral disease is less than a defined percentage.

SECONDARY OUTCOMES:
Development of methods and infrastructure for a national registry by recruiting participants from three distinct urban and rural regions within the UK (Norfolk, Leicestershire and London). | 1 year
  This will include an appraisal of a number of practical processes of recruitment, such as data acquisition, data processing and data management. This will inform future stages to expand the infrastructure to support a registry for widespread national use.
  More generally, the process of patient identification, recruitment, data collection and management will be the start of a much larger and broader national registry.
In conjunction with the Ménière's disease community, identify research questions which could be answered either using, or in collaboration with, a national registry. | through study completion, an average of 1 year
  In conjunction with the Ménière's disease community, identify research questions which could be answered either using, or in collaboration with, a national registry.

CONTACTS AND LOCATIONS:
Overall Officials: John Phillips, Consultant, Principal Investigator — Norfolk & Norwich University Hospitals NHS Foundation Trust
Locations (1):
- Norfolk & Norwich University Hospital, Norwich, Norfolk, United Kingdom